CLINICAL TRIAL: NCT00002796
Title: Phase I-II Study of Fluorouracil in Combination With Phenylbutyrate, Indomethacin and Recombinant Human Interferon-Gamma in Advanced Colorectal Cancer
Brief Title: Phase I-II Study of Fluorouracil in Combination With Phenylbutyrate in Advanced Colorectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00038; 96-322 ME*; CDR0000064879 (Registry Identifier: PDQ (Physician Data Query)); NCT01925326 (obsolete NCT alias)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Mucinous Adenocarcinoma of the Colon; Mucinous Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Signet Ring Adenocarcinoma of the Colon; Signet Ring Adenocarcinoma of the Rectum; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; 4-phenylbutyric acid; Indomethacin; Interferon-gamma; interferon gamma-1b

ARMS (1):
- Treatment (fluorouracil, phenylbutyrate, indomethacin, IFN-G (Experimental): Phase I: Patients receive 5-FU IV over 24 hours on day 1; phenylbutyrate IV over 120 hours and oral indomethacin daily on days 2-6; and interferon gamma subcutaneously on days 2, 4, and 6. Courses repeat weekly in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of 5-FU until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which less than 2 of 6 patients experience dose-limiting toxicity (DLT).
  Phase II: Patients receive 5-FU, phenylbutyrate, indomethacin, and interferon gamma as in phase I at the MTD.
  Interventions: Drug: fluorouracil; Drug: sodium phenylbutyrate; Drug: indomethacin; Biological: recombinant interferon gamma

INTERVENTIONS:
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: sodium phenylbutyrate — Given IV
  Other Names: Buphenyl; sodium 4-phenylbutyrate
Drug: indomethacin — Given orally
  Other Names: INDO; Indocin; Indometacin
Biological: recombinant interferon gamma — Given subcutaneously
  Other Names: Actimmune; gamma interferon; IFN-G

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Interferon-gamma may interfere with the growth of tumor cells and slow the growth of the tumor. Combining more than one drug with interferon-gamma may kill more tumor cells. This phase I/II trial is studying the side effects and best dose of giving fluorouracil together with phenylbutyrate, indomethacin, and interferon-gamma and to see how well it works in treating patients with stage IV colorectal cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine in a Phase I study the toxicity of flurouracil (FU) when given in escalating doses in combination with fixed doses of phenlylbutyrate (PB), indomethacin and recombinant human interferon-gamma (rhIFNg) to patients with advanced colorectal cancer.

II. To determine in a Phase II study the efficacy of FU in combination with PB, indomethacin and rhIFNg in patients with advanced colorectal cancer.

OUTLINE: This is a dose-escalation study of fluorouracil (5-FU).

Phase I: Patients receive 5-FU IV over 24 hours on day 1; phenylbutyrate IV over 120 hours and oral indomethacin daily on days 2-6; and interferon gamma subcutaneously on days 2, 4, and 6. Courses repeat weekly in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of 5-FU until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which less than 2 of 6 patients experience dose-limiting toxicity (DLT).

Phase II :Patients receive 5-FU, phenylbutyrate, indomethacin, and interferon gamma as in phase I at the MTD.

Patients are followed for survival.

PROJECTED ACCRUAL: A maximum of 24 patients will be accrued for the phase I portion of this study and approximately 46 patients will be accrued for the phase II portion of this study.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV colorectal adenocarcinoma, excluding brain metastases
* Histological confirmation of colorectal adenocarcinoma
* Previously untreated patients
* Previously treated patients

  * For the Phase I trial, no limitations
  * For the Phase II trial, previous treated limited to adjuvant radiation and/or chemotherapy which is completed at least 12 months before documentation of metastatic disease; patients may not have received chemotherapy for metastatic disease
* For the Phase I trial, patients may have measurable disease or unmeasurable disease; for the Phase II trial, patients must have measurable disease in at least two dimensions on x-rays, CT scan or MRI
* Expected survival of at least 16 weeks
* Performance status of >= 70% (Karnofsky)
* WBC >= 3000 uL
* Platelet count >= 100,000/uL
* Bilirubin =< 2 x ULN
* Creatinine =< 2 x ULN
* Not pregnant and not lactating; women of child bearing age must have negative pregnancy test (beta-hcg)
* No allergies to interferon-gamma or E.coli derived products
* No serious medical intercurrent medical illnesses, including Class III or IV cardiovascular disease; patient may not be dependent on immunosuppressive drugs including corticosteroids, and may not receive these drugs for the entire duration of the study
* No diarrhea, and with adequate oral intake
* Patients of child-bearing age and potential must agree to use adequate birth control other than oral contraceptives for the entire duration of the study
* No previous or concurrent malignancy except inactive nonmelanoma skin cancer, in situ carcinoma of the cervix, grade 1 bladder cancer, or other cancers if the patient has been disease free for >= 5 years
* Patients must be oriented and rational, and aware of the investigational nature of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1997-05; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Toxicity of flurouracil (FU) when given in escalating doses in combination with fixed doses of phenlylbutyrate (PB), indomethacin and recombinant human interferon-gamma (rhIFNg) to patients with advanced colorectal cancer (Phase I) | 1 week
Efficacy of FU in combination with PB, indomethacin and rhIFNg in patients with advanced colorectal cancer (Phase II) | Up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Max Sung, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States